CLINICAL TRIAL: NCT01409824
Title: Health Care Intervention Research-Quality of Prenatal and Maternal Care: Bridging the Know-do Gap (QUALMAT)
Brief Title: Health Care Intervention Research- Improving Pre-natal and Maternal Care
Acronym: QUALMAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: University Ghent (Other); Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Navrongo Health Research Centre, Ghana (Other); Karolinska Institutet (Other); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Prof. Rainer Sauerborn, University of Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: S-173/2008
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2010-02

CONDITIONS: Antenatal Care and Delivery
Keywords: clinical decision support system; performance based incentives; quality of maternal health care services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- without CDSS (No Intervention): This arm includes 6 health facilities in each partner country, where the clinical decision support system will not be implemented
  Interventions: Other: CDSS
- with CDSS (Experimental): This arm includes 6 health facilities in each partner country, where the clinical decision support system will be implemented, parallel to the performance based incentive package
  Interventions: Other: CDSS

INTERVENTIONS:
Other: CDSS — Clinical Decision Support System

SUMMARY:
Besides a dramatic lack of financial and human resources in developing countries, health care is additionally endangered by quality deficiencies caused by low staff motivation. This lack of motivation leads to an insufficient translation of knowledge into optimal utilization of resources. The "know-do" gap represents a challenge that must be addressed to strengthen health services performance towards achieving the Millennium Development Goals (MDGs). This is in particular true for some sensitive sectors like pre-natal and maternal health care. General objective of this research is to improve maternal health through better pre-natal and maternal care services offered by better motivated health workers. A computer-assisted clinical decision support system (CDSS) will be developed, implemented and tested aiming at (I) quality improvement of maternal and newborn care and (II) assessment of provider's performance. Based on this tool a commonly agreed incentive scheme to increase motivation will be shaped and tested in three SSA - countries, namely Burkina, Ghana, and Tanzania.

The incentive scheme might contain both non-monetary and monetary incentives and will be designed according to the human resource policy in the three countries. The planned approach is an implementation study with control arms containing one hospital and 6 first line health facilities in each of the study districts and an equal number of facilities in the control arm. A set of indicators for measurement of changes in quality of delivered services will be identified in order to follow up the sustainability and effectiveness of the strategies after their implementation. The study findings will allow understanding the important factors of staff motivation and facilitate adequate management for improvement of maternal and neonatal health care. "Knowing is not enough, we must apply; Wanting to do, is not enough, we must do it1"

- J.W. v. Goethe

ELIGIBILITY:
Inclusion Criteria:

* the patient in the primary health care center

Exclusion Criteria:

* patients outside the research regions

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
motivation | 2 years
  This research aims to increase the motivation of the health care providers through two parallel intervention packages- implementation of Clinical decision support system and incentive packages, based on the performance.

SECONDARY OUTCOMES:
Improved quality of health services in ANC and delivery | 2 years
  This research aims to improve the quality of the services provided through better motivated health workers

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Saronga HP, Duysburgh E, Massawe S, Dalaba MA, Wangwe P, Sukums F, Leshabari M, Blank A, Sauerborn R, Loukanova S. Cost-effectiveness of an electronic clinical decision support system for improving quality of antenatal and childbirth care in rural Tanzania: an intervention study. BMC Health Serv Res. 2017 Aug 7;17(1):537. doi: 10.1186/s12913-017-2457-z. PMID 28784130
- [Derived] Blank A, Prytherch H, Kaltschmidt J, Krings A, Sukums F, Mensah N, Zakane A, Loukanova S, Gustafsson LL, Sauerborn R, Haefeli WE. "Quality of prenatal and maternal care: bridging the know-do gap" (QUALMAT study): an electronic clinical decision support system for rural Sub-Saharan Africa. BMC Med Inform Decis Mak. 2013 Apr 10;13:44. doi: 10.1186/1472-6947-13-44. PMID 23574764
- See also: Improving pre-natal and maternal care — http://www.qualmat.net